CLINICAL TRIAL: NCT03408808
Title: Dorsal Wrist Ganglia; Aspiration Alone vs Aspiration and Injection of Platelet Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government); Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/091/17
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Ganglion of Wrist
Keywords: wrist; ganglion; platelet rich plasma; aspiration
MeSH Terms: conditions — Ganglion Cysts

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with two arms. Control - Aspiration alone. Intervention - aspiration plus injection of platelet righ plasma.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspiration alone (Active Comparator): The patients will have their dorsal wrist ganglion aspirated and then pressure dressing for 48 hours.
  Interventions: Procedure: Aspiration alone
- Aspiration plus platelet rich plasma (Experimental): The patients will have their dorsal wrist ganglion aspirated, and then injected with platelet rich plasma (derived from a blood sample taken at the same visit) and then pressure dressing for 48 hours.
  Interventions: Procedure: Platelet rich plasma

INTERVENTIONS:
Procedure: Platelet rich plasma — Aspiration of ganglion and injection with platelet rich plasma.
  Other Names: PRP
  Arms: Aspiration plus platelet rich plasma
Procedure: Aspiration alone — Aspiration of the ganglion
  Arms: Aspiration alone

SUMMARY:
Study to examine the efficacy of Platelet Rich Plasma (PRP) to reduce recurrence in dorsal wrist ganglia (DWG). We will compare aspiration alone and aspiration with injection of PRP.

We plan to recruit a maximum of 200 patients. We will assess the efficacy by contacting the patients by email or telephone at 6 weeks and 12 months. They will be asked to complete a questionnaire and a Patient Evaluated Measure score (PEMS). Adverse events will be screened for/ managed by a telephone call +/- review as necessary between 7 and 14 days.

DETAILED DESCRIPTION:
1. Patient selection All hand referrals vetted by Mr Lawrie or Miss Miller, those for dorsal wrist ganglia sent a letter of invitation and patient information. Patients responding to the letter with interested given an appointment at a special trial clinic.

   Contact details will be provided to allow any issues to be clarified discussed before attendance at clinic if the patient desires.
2. Assess eligibility/ enrolment in study - clinic visit 1

   1. All patients assessed by the chief investigator Mr David Lawrie (DFML) or Miss Katharine Hamlin (KH).
   2. Clinical assessment of presence of ganglion.
   3. Ensure not meeting exclusion criteria.
   4. If eligible and willing to complete study commitments discuss study and answer questions.
   5. Once we are happy the patient has understanding of the study and its risks then the patient will be asked if they wish to enrol or if they would like more time to consider.
   6. If they are willing to participate they will then be offered treatment in the same visit or a return visit
3. Intervention - clinic visit 1 or 2

   1. Check understanding and continuing desire to participate in study if 2nd visit.
   2. Complete consent form.
   3. Patient fills out a PEM score and demographics collected on SOS (Surgical Outcomes System - Arthrex).
   4. Randomisation.
   5. If in PRP group 15ml blood sample taken with Arthrex ACP double syringe and processed (see processing instructions in Appendix.9.
   6. Aspiration.
   7. If in PRP group - Injection of PRP (the same volume as aspirated).
   8. Pressure dressing with gauze, wool and crepe for 48 hours.
4. Adverse event screening/ management Patients are offered two options at the treatment visit.

1. Routine review at 10 - 14 days at the clinic or 2. Telephone review at 7 days by Miss Katharine Hamlin who will have performed the procedure.

On telephone review if the patient is entirely happy that there are no concerns then follow up will proceed by email or telephone as below.

If any concerns are raised, or if the patient desires, a face to face review will be arranged ideally within 24 hours but no longer than 72 hours. Recurrence or other outcomes will not be assessed at this time.

5. SOS/ Email/ Telephone interview - 1 (6 weeks)

a) Ganglion questionnaire b) PEM score c) Note any adverse events

6. SOS/ Email /Telephone interview - 2 (12 months)

1. Ganglion questionnaire
2. PEM score
3. Note any adverse events

ELIGIBILITY:
Inclusion Criteria:

* Solitary dorsal wrist ganglion.

Exclusion Criteria:

* Underlying wrist or ipsilateral arm pathology.
* Unable to consent to treatment.
* Unable or unwilling to attend follow up visits.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Hamlin, MBChB, Principal Investigator — NHS Grampian
Locations (1):
- NHS Grampian, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meena S, Gupta A. Dorsal wrist ganglion: Current review of literature. J Clin Orthop Trauma. 2014 Jun;5(2):59-64. doi: 10.1016/j.jcot.2014.01.006. Epub 2014 Jun 3. PMID 25983472 (Retraction: PMID 34589409 J Clin Orthop Trauma. 2020 Sep 17;11(Suppl 5):S916)
- [Background] Janzon L, Niechajev IA. Wrist ganglia. Incidence and recurrence rate after operation. Scand J Plast Reconstr Surg. 1981;15(1):53-6. doi: 10.3109/02844318109103412. PMID 7268314
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Freymiller EG, Aghaloo TL. Platelet-rich plasma: ready or not? J Oral Maxillofac Surg. 2004 Apr;62(4):484-8. doi: 10.1016/j.joms.2003.08.021. No abstract available. PMID 15085518
- [Background] Yu W, Wang J, Yin J. Platelet-rich plasma: a promising product for treatment of peripheral nerve regeneration after nerve injury. Int J Neurosci. 2011 Apr;121(4):176-80. doi: 10.3109/00207454.2010.544432. Epub 2011 Jan 19. PMID 21244302
- [Background] Valente Duarte de Sousa IC, Tosti A. New investigational drugs for androgenetic alopecia. Expert Opin Investig Drugs. 2013 May;22(5):573-89. doi: 10.1517/13543784.2013.784743. Epub 2013 Apr 4. PMID 23550739
- [Background] Marx RE. Platelet-rich plasma (PRP): what is PRP and what is not PRP? Implant Dent. 2001;10(4):225-8. doi: 10.1097/00008505-200110000-00002. No abstract available. PMID 11813662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma
Started | 8 | 9
Completed | 8 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: years] | 33.9 [23 to 46] | 23.2 [18 to 29] | 28.6 [18 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Recurrence of Ganglia
Description: Has the ganglion returned?
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma
Number analyzed (Participants) | 8 | 8
Participants | 8 | 5

2. Primary Outcome: Number of Participants With a Recurrence of Ganglia
Description: Has the ganglion returned?
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma
Number analyzed (Participants) | 8 | 8
Participants | 3 | 7

3. Secondary Outcome: PEM Score
Description: The Patient Evaluation Measure (PEM) (Macey and Burke, 1995) is used to measure outcomes in hand surgery. It consists of a series of 18 questions, which address different aspects of symptoms pertaining to the hand and hand function. The questions have been split into three sections, the first being five questions on treatment. The second section contains ten questions on the condition of your hand at this moment in time (Feeling, Cold intolerance, Pain, Dexterity, Movement, Grip, ADL, Work, Appearance and Hand in general) and the third section is an overall assessment containing three questions. Each question from sections two and three are marked from 1-7, 7 being the worst outcome and 1 being the best outcome. The answers are expressed as a percentage disability ranging from zero to 100, with lower scores indicating less disability and are therefore better. This questionnaire is reliable, valid and responsive for assessing wrist disorders (Dias et al., 2001).
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma
Number analyzed (Participants) | 8 | 8
score on a scale | 40.2 [27.8 to 58.6] | 38.7 [15.8 to 66.9]

4. Secondary Outcome: PEM Score
Description: as for outcome 3
Time Frame: 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma
Number analyzed (Participants) | 8 | 8
score on a scale | 35 [14.3 to 66.2] | 40.6 [14.3 to 57.1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Aspiration Alone | Aspiration Plus Platelet Rich Plasma
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03408808/Prot_SAP_003.pdf
  • Informed Consent Form (2018-06-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03408808/ICF_002.pdf